CLINICAL TRIAL: NCT01342198
Title: A Phase 1, Open-Label, Randomized, Cross-Over Study to Evaluate the Effects of Multiple Doses of Erythromycin on the Pharmacokinetics of a Single Dose of Pregabalin Controlled Release in Healthy Subjects
Brief Title: An Investigation of the Effects of Erythromycin on the Pharmacokinetics of the Pregabalin Controlled Release Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A0081197
Record Dates: First submitted 2011-04-21; First posted 2011-04-27 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2011-07

CONDITIONS: Healthy
Keywords: pregabalin; pharmacokinetics; bioavailability; bioequivalence
MeSH Terms: interventions — Erythromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Single Dose Pregabalin Controlled Release
  Interventions: Drug: Pregabalin controlled release, 330 mg
- 2 (Experimental): Single Dose Pregabalin Controlled Release with Multiple Doses of Erythromycin
  Interventions: Drug: Pregabalin controlled release, 330 mg; Drug: erythromycin

INTERVENTIONS:
Drug: Pregabalin controlled release, 330 mg — A single oral dose of 330 mg controlled release tablet
  Arms: 1
Drug: Pregabalin controlled release, 330 mg — A single oral dose of 330 mg controlled release tablet
  Arms: 2
Drug: erythromycin — A total of three doses of 500 mg erythromycin ethylsuccinate tablets administered six hours apart beginning approximately 1 hour prior to pregabalin CR
  Arms: 2

SUMMARY:
The purpose of this study is to 1) evaluate the extent of absorption of a single dose of a pregabalin controlled release tablet with and without coadministration of erythromycin and 2) evaluate the safety and tolerability of a single dose of a pregabalin controlled release tablet with and without coadministration of erythromycin.

DETAILED DESCRIPTION:
Evaluate the absorption, pharmacokinetics, safety/tolerability of a single dose of a pregabalin CR tablet with and without erythromycin

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or females
* Between the ages of 18 and 55 years, inclusive
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2

Exclusion Criteria:

* Illicit drug use
* Pregnant or nursing females
* Females of childbearing potential who are unwilling or unable to use an acceptable method of contraception

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Area under the curve from 0 to infinity (AUCinf) | 3 days
Peak concentrations (Cmax) for assessment of equivalence between controlled released (CR) alone and CR with erythromycin | 3 days

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081197&StudyName=An%20Investigation%20of%20the%20Effects%20of%20Erythromycin%20on%20the%20Pharmacokinetics%20of%20the%20Pregabalin%20Controlled%20Release%20Tablet